CLINICAL TRIAL: NCT06451302
Title: A Prospective Multicenter Cohort Study of Outcome and Safety Profile of Risk Stratification Oriented Treatment in Pediatric Ewing Sarcoma in China
Brief Title: Risk Stratification Oriented Treatment of Pediatric Ewing Sarcoma: a Prospective Multicenter Cohort Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-Ewing sarcoma
Record Dates: First submitted 2024-06-02; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Ewing Sarcoma; Risk Stratification
Keywords: risk-stratified treatment
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Cyclophosphamide; Doxorubicin; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Description: Participants receive the straified treatment according to assigned risk group (Experimental): Patients with Ewing sarcoma are risk stratified according to definition. Patients with low risk receive 8 cycles of chemotherapy comprising low-dose cyclosphomide, adriamycin，vincristine(CAV) alternated with ifosfamide and etoposide(IE). Patients with moderate risk receive a total of 12 cycles of moderate-dose CAV and IE. Patients with high risk receive a total of 17 cycles of high-dose CAV and IE. Thereafter, maitenance therapy is administered to high-risk patients after chemotherapy.
  Interventions: Drug: cyclophosphamide, adriamycin, vincristine，Ifosfamide，etoposide

INTERVENTIONS:
Drug: cyclophosphamide, adriamycin, vincristine，Ifosfamide，etoposide — The doses and intensity of chemotherapy vary according to risk stratification. Mainenance therapy is added to high-risk patients.
  Other Names: vinorelbine

SUMMARY:
The aim is to evaluate the outcome and safety of risk-stratification oriented treatment for pediatric Ewing sarcoma in multicenters .

DETAILED DESCRIPTION:
Pediatric Ewing sarcoma is stratified into three risk groups(low risk, moderate risk and high risk) accordiong to age, longest diameter of lesion, volume and tumor site. Participants receive chemotherapy with corresponding intensity. The prospective study is to assess efficacy, outcome and safety profile of different treatment received for pediatric Ewing sarcoma.

The prospecitive single-arm study is to be conducted in Chinese multicenters.

ELIGIBILITY:
Inclusion Criteria:

* age≤18 years, no gender limitation;
* The ECOG （performance status，PS）is 0～1 score;
* The expected survival time is not less than 12 weeks;
* Heart function: A) Cardiac COLOR ultrasound detection LVEF≥ 50%; B) EKG suggests no myocardial ischemia;C) No history of arrhythmia requiring drug intervention before enrollment;
* Patients who meet the clinical diagnostic criteria and are diagnosed with pediatric Ewing sarcoma;
* Patients who have progressed, relapsed or refractory after first-line treatment (failed to achieve complete or partial response after recent treatment);
* Measurable lesions (according to RECIST 1.1 standards, CT scan length of tumor lesions ≥10mm, CT scan short diameter of lymph node lesions ≥15mm, measurable lesions have not received radiotherapy, freezing and other local treatments);
* The patient must fully recover from the acute toxic effects of all previous anticancer chemotherapy: A) Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (42 days if nitrosourea was used previously);B) Experimental drug or anticancer therapy other than chemotherapy: not available within the first 28 days of planned initiation of AI or VIT. Complete recovery from clinically significant toxicity of the therapy must be determined;C) Hematopoietic growth factor: at least 14 days after the last administration of long-acting growth factor or 3 days after the last administration of short-acting growth factor;D) Immunotherapy: at least 42 days after completion of any type of immunotherapy (except steroids), such as immune checkpoint inhibitors and tumor vaccines; E) X-ray therapy (XRT) : at least 14 days after local palliative XRT (small mouth); For other substantial bone marrow (BM) irradiation, it must be completed for at least 42 days; F) Stem cell infusion without total body irradiation (TBI) : there is no evidence of active graft-versus-host disease and the transplant or stem cell infusion must be completed at least 56 days after the infusion;
* Laboratory tests during screening should meet the following conditions: A) Absolute value of neutrophils (ANC) ≥1.5×109/L (if bone marrow invasion, ANC≥1.0×109/L); B) Platelet count (PLT) ≥75×109/L (PLT≥50×109/L for bone marrow invasion); C) Bilirubin (sum of combined + uncombined) ≤ 2.5× upper limit of normal value (ULN) (corresponding to age), patients with confirmed Gilbert's syndrome can be included in the group according to the investigator's judgment; D) Estimated glomerular filtration rate ≥30 mL/min/1.73 m2 or serum creatinine (Cr) ≤ 1.5ULN (calculated according to the standard Cockcroft-Gault formula); E) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN (5 times ULN if liver metastasis is present)
* Able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits during the study period;
* The parent/guardian of the child or adolescent subject is capable of understanding, agreeing to, and signing the study Informed consent (ICF) and the applicable child consent form prior to initiating any program-related procedures; Subject is capable of expressing consent with parental/guardian consent (if applicable).

Exclusion Criteria:

* Exclusion criteria

  * Patients who have symptomatic brain metastasis except that who completed therapy 21 days prior to enrollment and had stable disease related to brain metastasis confirmed by cerebral CT or MRI or radiography;
  * Previous or concurrent clinical significance of active cardiovascular diseases, including congenital heart disease or pericardial disease, history of heart failure, myocardial infarction, coronary heart disease, heart valvular disease, cardiomyopathy, arrhythmias (including persistent atrial fibrillation, complete left bundle branch block, frequent ventricular premature onset); Or prolonged QT interval (QTc) after current corrected heart rate > 480 ms; Patients with grade III ~ IV cardiac insufficiency according to the New York Heart Association (NYHA) cardiac function classification (age > 3 years) or infant cardiac function standard (age ≤3 years), or left ventricular ejection fraction (LVEF) < 50% as indicated by color doppler echocardiography;
  * Patients with a history of pulmonary interstitial disease or concurrent pulmonary interstitial disease;
  * Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), with a tendency to bleed or undergoing thrombolytic or anticoagulant treatment;
  * Severe chronic skin diseases in the past;
  * Previous allergic asthma or severe allergic disease;
  * Poorly controlled hypertension and diabetes;
  * Have a history of other tumors;
  * HIV or syphilis infected patients;
  * Patients who have previously received organ transplants;
  * Uncontrolled and active systemic bacterial, viral or fungal infection;
  * Contraindications to the use of large doses of hormones, such as uncontrolled hyperglycemia, gastric ulcers or mental diseases;
  * Have a history of severe neurological or psychiatric disorders, including epilepsy or autism.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | from initial diagnosis to 5 years after EOT
  The proportion of patients who achieved CR or PR

SECONDARY OUTCOMES:
OS | from start of treatment to 5 years after EOT
  The time from from start of treatment to death or loss of follow-up
EFS | from start of treatment to 5 years after EOT
  The time from from start of treatment to disease progression, recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No